CLINICAL TRIAL: NCT07398963
Title: Exploratory Study of Oncolytic Vaccinia VIrus-Delivered Targeted CD19 In Vivo CAR-T/M Therapy for Refractory/Relapsed B-Cell Lymphoma
Brief Title: Clinical Study of Oncolytic Vaccinia VIrus Delivering Targeted CD19 in Vivo CAR-T/M Therapy for Refractory/Relapsed B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2026-0013
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Refractory/Relapsed B-cell Lymphoma
Keywords: Oncolytic poxvirus; In vivo CAR-T
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intratumoral or intravenous injection RGV005 (Experimental): Subjects will receive intratumoral injections of CD19-CAR oncolytic vaccinia virus (RGV005)
  Interventions: Biological: CD19-CAR novel oncolytic vaccinia virus

INTERVENTIONS:
Biological: CD19-CAR novel oncolytic vaccinia virus — Injection of CD19-CAR novel oncolytic vaccinia virus which carrying the CD19-CAR gene (RGV005) is designed to locally induce the in situ generation of CAR-T and CAR-M cells in tumors for precise lymphoma killing.

SUMMARY:
To study the safety and effectiveness of oncolytic Vaccinia VIrus-Delivered Targeted CD19 In Vivo CAR-T/M Therapy for Refractory/Relapsed B-Cell Lymphoma

DETAILED DESCRIPTION:
This is a single-arm, dose-escalation, non-randomized, multicenter, dose-escalation exploratory study aimed at evaluating the safety and efficacy of a novel CD19-CAR oncolytic vaccinia virus (RGV005) in patients with B-cell lymphoma.

The study included two groups: (1) intratumoral injection group (12-24 patients); (2) intravenous injection group (12-24 patients). A standard 3×3 design will be used to conduct a single-dose escalation safety and tolerability trial. Patients will be assigned to one of four dose groups in ascending order: Dose Group 1 (1×10^8 pfu), Dose Group 2 (3×10^8 pfu), Dose Group 3 (1×10^9 pfu), and Dose Group 4 (3×10^9 pfu). Each dose group plans to recruit 3 subjects. After completing the treatment and the month-3 assessment visit, subjects will enter the long-term follow-up period, which will last for 3 years after administration for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old, up to 75 years old, male or female;
2. ECOG score 0-2;
3. Histologically confirmed non-Hodgkin B-cell lymphoma (NHL) [diagnostic criteria are WHO2008], including diffuse large B-cell lymphoma (DLBCL) non-specific, primary mediastinal large B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL), transformed follicular cell lymphoma (TFL) and other indolent B-cell NHL transformed types;
4. CD19 positive (immunohistochemistry or flow cytometry);
5. DLBCL refractory or relapse is defined as: complete remission after 2 lines of therapy; Disease progression during any course of treatment, or disease stabilization time equal to and less than 6 months; or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation;
6. MCL: Complete remission after 2 lines of treatment (including BTK inhibitors); Disease progression during any course of treatment, or disease stabilization time equal to and less than 6 months; or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation;
7. At least one measurable superficial lesion, requiring any length diameter of lymph node lesion greater than 1.5cm or any length diameter of extranodal lesion greater than 1.0cm, and uptake of the lesion on PET-CT scan (SUV greater than hepatic blood pool);
8. Absolute peripheral blood neutrophil ≥ 1000/mm3, platelet ≥ 50,000/mm3;
9. Heart, liver and kidney function: creatinine <1.5mg/dL; ALT (alanine aminotransferase)/AST (aspartate aminotransferase) less than 2.5 times the upper limit of normal; Total bilirubin < 1.5 mg/dL; Cardiac ejection fraction (EF) ≥ 50%;
10. Have sufficient understanding ability and voluntarily sign the informed consent form;
11. Women of childbearing potential must have a negative serum pregnancy test and agree to practice effective birth control during the treatment phase and for 60 days after the last application of oncolytic virus;
12. Male patients must agree to practice effective birth control during the study and for 60 days after the last viral treatment.

Exclusion Criteria:

1. History of other tumors;
2. Vaccination with the smallpox vaccine within 3 months before or during the study treatment;
3. Receiving gene therapy or any type of oncolytic virus therapy within 3 months before the study treatment;
4. Other open wounds;
5. Active autoimmune diseases;
6. Uncontrolled active infections;
7. HIV infection, uncontrolled HBV, HCV, or syphilis infection;
8. Known central nervous system lymphoma;
9. Clinically significant heart disease;
10. Allergy to albumin or egg products;
11. History of organ transplantation or similar surgeries;
12. Need for systemic treatment for skin diseases;
13. History of severe systemic reactions or side effects after smallpox vaccination;
14. Known alcohol or viral dependence;
15. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety, and tolerability, and determine the recommended dosage of the CD19-CAR novel oncolytic vaccinia virus

SECONDARY OUTCOMES:
Complete response rate (CR) | Up to 2 years
  To determine the anti-tumor effectivity of To determine the anti-tumor effectivity of the CD19-CAR novel oncolytic vaccinia virus
Progression free survival (PFS) | Up to 2 years
Duration of response (DOR) | Up to 2 years
Overall survival (OS) | Up to 2 years
Partial response rate (PR) | Up to 2 years
Overall response rate (ORR) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No